CLINICAL TRIAL: NCT03699761
Title: Evaluation of Pelvic Peritonization in Robotic or Laparoscopic Low Anterior Resection for Rectal Cancer
Brief Title: The Role of Pelvic Peritonization in Laparoscopic or Robotic Low Anterior Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Tang Bo, Principal Investigator, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POLAR
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Rectum Cancer
Keywords: Anastomotic leakage; Complication; Reoperation; Pelvic Peritonization
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Peritonization (Experimental)
  Interventions: Procedure: Closure of the pelvic peritoneum; Procedure: Nonclosure of the pelvic peritoneum
- Without Pelvic Peritonization (No Intervention)

INTERVENTIONS:
Procedure: Closure of the pelvic peritoneum — Closure of the pelvic peritoneum after anastomosis for middle-low rectal caner.
  Arms: Pelvic Peritonization
Procedure: Nonclosure of the pelvic peritoneum — Nonclosure of the pelvic peritoneum after anastomosis for middle-low rectal caner.
  Arms: Pelvic Peritonization

SUMMARY:
A randomized controlled clinical trial to compare the short and long outcomes of low anterior resection for middle-low rectal cancer with or without pelvic peritonization.

ELIGIBILITY:
Inclusion Criteria:

* Matching the diagnostic criteria of rectal adenocarcinoma
* Laparoscopic or robotic radical surgery for rectal cancer
* Preoperative TNM staging T1-3N0-2M0
* No history of malignant tumors by preoperative examination
* Middle and low rectal cancer
* Tumor size of 4 cm or less
* ASA 1-3 scores
* Written informed consent by the patient
* The patient is willing to randomize to any group

Exclusion Criteria:

* Previous abdominal surgery
* Past malignant tumor history
* Preoperative examination suggests distant metastasis
* Be participating or have participated in other clinical studies related to rectal cancer surgery within 6 months
* Emergency operation

Elimination criteria

* The tumor is confirmed to be T4b during the operation or other tumors are found to be combined with other tumors during the operation
* The anastomosis is located above the peritoneum reflex
* Intraoperative conversion to laparotomy
* Change the surgical method to perform Miles or Hartmann surgery
* Postoperative pathologically confirmed non-adenocarcinoma
* The patient asked to withdraw

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Grade III-IV complications | 30 days
  The rate of grade III-IV complication according to Clavien-Dindo classification after low anterior resection

SECONDARY OUTCOMES:
Rate of reoperation | 30 days
  The rate of reoperation after leakage
Detection of inflammation markers | 7 days
  C-reactive protein(1, 3, 5, 7 days after operation, and 1 day before discharge, all blood drawn is venous blood)
The rate of anastomotic leakage | 30 days
  Clinical diagnostic criteria for anastomotic leakage: 1. Abdominal and systemic infection symptoms: abdominal pain, bloating, fever, elevated white blood cells, PCT, CRP and other inflammation indicators; 2. Gas, pus, feces passing through the pelvic drainage tube, abdominal incision, etc.
Hospital time | 30 days
  Comparison of hospital stay between the two groups
Overall complication rate | 30days
  Overall complication rate include I-IV grade
Estimated blood loss | 1 day
  Blood loss will be measured according to the suction and the weight of wet gauze, and then minus the irrigation
Operation time | 1 day
  The time from start to end of surgery
Postoperative bleeding | 7 days
  Postoperative intra-abdominal bleeding
Intestinal obstruction | 30 days
  Incidence of intestinal obstruction caused by various reasons after surgery
Readmission rate | 30 days
  Rate of hospital readmissions due to complications after discharge
LARS | 12 months
  Low Anterior resection syndrome caused by rectal surgery
Acute inflammatory Response | 7 days
  Procalcitonin(1, 3, 5, 7 days after operation, and 1 day before discharge, all blood drawn is venous blood)
Acute inflammatory Response | 7 days
  Check Neutrophils(1, 3, 5, 7 days after operation, and 1 day before discharge, all blood drawn is venous blood)
Detection of other inflammation markers | 7 days
  interleukin-6(1, 3, 5, 7 days after operation, and 1 day before discharge, all blood drawn is venous blood)
Treatment cost | 30 days
  Comparison of cost between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- General Surgery Center of PLA, Chongqing, China